CLINICAL TRIAL: NCT03224507
Title: Monoclonal Antibody-Based Sequential Therapy for Deep Remission in Multiple Myeloma - MASTER Trial
Brief Title: Monoclonal Antibody-Based Sequential Therapy for Deep Remission in Multiple Myeloma
Acronym: MASTER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Amgen (Industry); Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Luciano Jose Costa, MD, Associate Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: F170525008 (UAB 1735)
Record Dates: First submitted 2017-07-10; First posted 2017-07-21 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; induction therapy; autologous hematopoietic cell transplantation; KRdD; Daratumumab; Carfilzomib; Lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Lenalidomide; Dexamethasone; daratumumab

STUDY DESIGN:
Intervention Model Description: The study has four cycles (28-days each) of drug therapy prior to being evaluated for auto-HCT. After the completion of induction therapy, the patient will be evaluated for a transplant of their own hematopoietic stem cells. If, after the transplant, the patient still has detectable multiple myeloma, the patient will proceed to a series of consolidation blocks, up to three, consisting of four cycles of the KRdD at specified dosages and time frames. After completion of consolidation therapy, maintenance therapy will begin until disease progression or intolerance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KRdD followed by auto-HCT (Experimental): Cycle 1-Dexamethasone 40mg orally days 1/8/15/22; Lenalidomide 25mg orally days 1-21; Carfilzomib 20mg/m2 days 8/9 then 36mg/m2 venous days 15/16; Daratumumab 16mg/kg venous days 1/8/15/22 (KRd-Dara). Cycle 2 the same except Carfilzomib 36mg/m2 venous days 1/2/8/9/15/16. Cycles 3,4 the same but no Daratumumab Days 8 and 22. Dosage adjusted for last tolerated dose (LTD). Following induction therapy, auto-HCT is done (consolidation 1), then up to two 4-cycle blocks of KRd-Dara consolidation (consolidations 2 and 3). Minimum residual disease (MRD) checked after each phase. Patients with confirmed MRD(-) at or after consolidation 1 will not undergo maintenance and will be actively monitored for resurgence of MRD or clinical relapse. After consolidation if MRD+ patients will undergo standard of care lenalidomide maintenance.
  Interventions: Drug: KRdD followed by auto-HCT
- KRdD only (Experimental): Cycle 1-Dexamethasone 40mg orally days 1/8/15/22; Lenalidomide 25mg orally days 1-21; Carfilzomib 20mg/m2 days 8/9 then @ 36mg/m2 venous days 15/16; Daratumumab 16mg/kg venous days 1/8/15/22. Cycle 2 the same except Carfilzomib 36mg/m2 venous days 1/2/8/9/15/16. Cycles 3,4 the same but no Daratumumab Day 22. Dosage adjusted for last tolerated dose (LTD). Following induction therapy, Following induction therapy, patients will receive up to three 4-cycle blocks of KRd-Dara consolidation (consolidations 1, 2 and 3). Minimum residual disease (MRD) checked after each phase. Patients with confirmed MRD(-) at or after consolidation 1 will not undergo maintenance and will be actively monitored for resurgence of MRD or clinical relapse. After consolidation if MRD+ patients will undergo standard of care lenalidomide maintenance.
  Interventions: Drug: KRdD only

INTERVENTIONS:
Drug: KRdD followed by auto-HCT — Dosages of each drug will vary depending on therapy type and cycle number. KRdD therapy will be followed by autologous hematopoietic cell transplantation and KRdD consolidation.
  Other Names: KRdD = Kyprolis (Carfilzomib), Revlimid (Lenalidomide), dexamethasone, Darzalex (Daratumumab)
  Arms: KRdD followed by auto-HCT
Drug: KRdD only — Dosages of each drug will vary depending on therapy type and cycle number. KRdD therapy will not be followed by autologous hematopoietic cell transplantation but will proceed with KRdD consolidation.
  Other Names: KRdD = Kyprolis (Carfilzomib), Revlimid (Lenalidomide), dexamethasone, Darzalex (Daratumumab)
  Arms: KRdD only

SUMMARY:
Multiple myeloma (MM), a plasma cell disorder, is the second most common hematologic malignancy in the U.S. No standard curative therapy has yet been found. A variety of therapeutic measures including high dose melphalan, induction therapy, and continuous therapy have been used but the goal of complete response without relapse has not been achieved. More active treatment regimens and better tools for response assessment are needed.

DETAILED DESCRIPTION:
This trial will assess the safety and efficacy of an induction therapy using the combination of dexamethasone, lenalidomide (revlimid), daratumumab (Darzalex) and carfilzomib (Kyprolis) to treat patients with newly diagnosed multiple myeloma. The therapy with KRdD (Kyprolis, Revlimid, dexamethasone, Darzalex) will be followed by autologous hematopoietic cell transplantation (auto-HCT) and KRdD consolidation. Duration of therapy will be guided by eradication of minimal residual disease (MRD). The hypothesis is that the KRdD therapy particularly in combination with the auto-HCT will be safe and lead to deep remission. Patients who become MRD- will discontinue therapy (no maintenance therapy) and be actively monitored for resurgence of MRD or clinical relapse.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years with no upper age limit
* Diagnosis of newly diagnosed multiple myeloma with indication for initiation of therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* No prior MM-directed therapy except for dexamethasone (up to 160 mg) and/or bortezomib (up to 5.2 mg/m2) and/or cyclophosphamide up to 1000 mg/m2 administered for management of acute manifestations of MM (hypercalcemia, renal impairment, pain) for no longer than 4 weeks prior to enrollment. If subject received any prior therapy, pretreatment parameters necessary for disease characterization and response assessment must be available.
* Measurable disease meeting at least one of the following criteria:

  1. Serum monoclonal (M) protein ≥1.0 g/dl
  2. ≥ 200 mg of M protein/24h in the urine
  3. Serum-free light chain ≥10 mg/dL and abnormal kappa to lambda ratio.
* Life expectancy ≥12 months.
* Adequate hepatic function, with serum ALT ≤ 3.5 times the upper limit of normal and serum direct bilirubin ≤ 2 mg/dL (34 μmol/L) within 21 days prior to initiation of therapy.
* Creatinine clearance (CrCl) ≥ 40 mL/minute within 21 days prior to start of therapy either measured or calculated using a standard formula (eg. Cockcroft and Gault).
* Written informed consent in accordance with federal, local, and institutional guidelines.
* Females of childbearing potential must agree to ongoing pregnancy testing and to practice contraception. Male subjects must agree to practice contraception.
* All subjects must agree to comply with and be enrolled in Revlimid REMS program.

Exclusion Criteria:

* Diagnosis of amyloidosis, Crow-Fukase syndrome, Waldenstrom's macroglobulinemia, smoldering MM.
* Major surgery, radiotherapy or infection requiring therapy within 14 days of starting treatment.
* Known FEV1 or cDLCO < 50% of predicted.
* Pregnant or lactating females.
* Known human immunodeficiency virus infection.
* Active hepatitis B (Hepatitis B core antibody positive and subsequent Hepatitis B surface antigen positive or Hepatitis B DNA positive) or C infection (Hepatitis C antibody positive and subsequent detectable viral load).
* Unstable angina or myocardial infarction within 4 months prior to registration, New York Heart Association Class II, III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker.
* Cerebrovascular disease manifested as prior stroke at any time or TIA in the 12 months prior to initiation of therapy
* Non-hematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or localized thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas.
* Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 21 days prior to registration.
* Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib).
* Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 21 days prior to registration.
* Contraindication or intolerance to required supportive care medications (Aspirin and Acyclovir).
* Any other clinically significant medical disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luciano J Costa, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - University of Wisconsin, school of medicine and public health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giri S, Dhakal B, Callander NS, Medvedova E, Godby K, Dholaria BR, Bal S, Ravi G, Chhabra S, Silbermann RW, Costa L. Optimal MRD-based end point to support response-adapted treatment cessation in newly diagnosed multiple myeloma. Blood. 2025 Aug 7;146(6):707-716. doi: 10.1182/blood.2024027674. PMID 40193714
- [Derived] Callander NS, Silbermann R, Kaufman JL, Godby KN, Laubach J, Schmidt TM, Sborov DW, Medvedova E, Reeves B, Dhakal B, Rodriguez C, Chhabra S, Chari A, Bal S, Anderson LD Jr, Dholaria BR, Nathwani N, Hari P, Shah N, Bumma N, Holstein SA, Costello C, Jakubowiak A, Wildes TM, Orlowski RZ, Shain KH, Cowan AJ, Pei H, Cortoos A, Patel S, Lin TS, Giri S, Costa LJ, Usmani SZ, Richardson PG, Voorhees PM. Daratumumab-based quadruplet therapy for transplant-eligible newly diagnosed multiple myeloma with high cytogenetic risk. Blood Cancer J. 2024 Apr 22;14(1):69. doi: 10.1038/s41408-024-01030-w. PMID 38649340
- [Derived] Costa LJ, Chhabra S, Medvedova E, Dholaria BR, Schmidt TM, Godby KN, Silbermann R, Dhakal B, Bal S, Giri S, D'Souza A, Hall AC, Hardwick P, Omel J, Cornell RF, Hari P, Callander NS. Minimal residual disease response-adapted therapy in newly diagnosed multiple myeloma (MASTER): final report of the multicentre, single-arm, phase 2 trial. Lancet Haematol. 2023 Nov;10(11):e890-e901. doi: 10.1016/S2352-3026(23)00236-3. Epub 2023 Sep 27. PMID 37776872
- [Derived] Costa LJ, Chhabra S, Medvedova E, Dholaria BR, Schmidt TM, Godby KN, Silbermann R, Dhakal B, Bal S, Giri S, D'Souza A, Hall A, Hardwick P, Omel J, Cornell RF, Hari P, Callander NS. Daratumumab, Carfilzomib, Lenalidomide, and Dexamethasone With Minimal Residual Disease Response-Adapted Therapy in Newly Diagnosed Multiple Myeloma. J Clin Oncol. 2022 Sep 1;40(25):2901-2912. doi: 10.1200/JCO.21.01935. Epub 2021 Dec 13. PMID 34898239

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There was no randomization between KRdD followed by Auto-HCT and KRdD alone. Assignment was per suitability for ASCT. In the end all participants were considered suitable for ASCT, hence the enrollment of zero patients in the KRdD arm
Period: Overall Study
Arm/Group | KRdD Followed by Auto-HCT | KRdD Only
Started | 123 | 0
Completed | 108 | 0
Not Completed | 15 | 0
Not completed — Death | 3 | 0
Not completed — Lack of Efficacy | 6 | 0
Not completed — Withdrawal by Subject | 6 | 0

BASELINE CHARACTERISTICS:
Population: All enrolling patients
Groups:
- Total: Total of all reporting groups
Arm/Group | KRdD Followed by Auto-HCT | KRdD Only | Total
Number analyzed (Participants) | 123 | 0 | 123
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [55 to 68] |  | 61 [55 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 |  | 53
  Male | 70 |  | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 2 |  | 2
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 25 |  | 25
  White | 94 |  | 94
  More than one race | 2 |  | 2
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 123 |  | 123

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With MRD(-) Remissions at the Completion of Consolidation Therapy
Description: The primary endpoint of MRD(-) rate, or percentage of patients with MRD(-) remissions, will be estimated along with two-sided 95% confidence interval using Clopper-Pearson exact method. Simon's optimal two-stage design will be utilized in determining the rate of MRD(-) cases. MRD assessment will be done with ClonoSEQ to identify myeloma-specific sequences.
Time Frame: Baseline until MRD(-) is reached estimated to be up to 15 months.
Population: Patients with trackable clonogenic sequence by NGS
Measure: Number (95% Confidence Interval); unit: percentage of patients achieving MRD (-)
Arm/Group | KRdD Followed by Auto-HCT | KRdD Only
Number analyzed (Participants) | 118 | 0
percentage of patients achieving MRD (-) | 81.4 [73.1 to 87.9] |

2. Secondary Outcome: Serious Adverse Events (SAEs) From the KRdD Treatment
Description: The Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be used for this assessment. SAEs include events that are Grade 3 and above; non-serious events are Grades 1-2.
Time Frame: Baseline until the progression of disease or MRD(-) status up to an estimated 15 months.
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | KRdD Followed by Auto-HCT | KRdD Only
Number analyzed (Participants) | 123 | 0
Participants | 14 |

3. Secondary Outcome: Percentage of Patients With MRD(-) Status at the Completion of Induction Therapy
Description: The primary endpoint of MRD(-) rate will be estimated along with two-sided 95% confidence interval using Clopper-Pearson exact method. Simon's optimal two-stage design will be utilized in determining the rate of MRD(-) cases. MRD assessment will be done with ClonoSEQ to identify myeloma-specific sequences.
Time Frame: Baseline until MRD(-) status estimated at 6 months or until disease progression
Population: All participants with trackable clonogenic sequences by NGS
Measure: Count of Participants; unit: Participants
Arm/Group | KRdD Followed by Auto-HCT | KRdD Only
Number analyzed (Participants) | 118 | 0
Participants | 45 |

4. Secondary Outcome: Percentage of Patients With Auto-HCT That Convert From Positive to Negative MRD
Description: as for outcome 3
Time Frame: From baseline up to an estimated 9 months
Population: Patients with clonogenic sequence and MRD>= 10-5 post induction
Measure: Count of Participants; unit: Participants
Arm/Group | KRdD Followed by Auto-HCT | KRdD Only
Number analyzed (Participants) | 73 | 0
Participants | 32 |

5. Secondary Outcome: Percentage of Patients Achieving Complete Remission Following Complete Therapy
Description: The primary endpoint of MRD(-) rate will be estimated along with two-sided 95% confidence interval using Clopper-Pearson exact method. Simon's optimal two-stage design will be utilized in determining the rate of MRD(-) cases. MRD assessment will be done with ClonoSEQ to identify myeloma-specific sequences. Complete therapy incorporates induction and consolidation therapy.
Time Frame: Baseline up to 15 months
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | KRdD Followed by Auto-HCT | KRdD Only
Number analyzed (Participants) | 123 | 0
Participants | 106 |

6. Secondary Outcome: Percentage of Patients That Convert From MRD(-) to MRD(+) Following Treatment Discontinuation
Description: as for outcome 3
Time Frame: Baseline to 2 years
Population: All patients with confirmed MRD negativity transitioning to observation
Measure: Count of Participants; unit: Participants
Arm/Group | KRdD Followed by Auto-HCT | KRdD Only
Number analyzed (Participants) | 84 | 0
Participants | 23 |

7. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the interval from the start of therapy to the earliest occurrence of the following: disease progression, initiation of anti-myeloma therapy that is not an accepted maintenance therapy of lenalidomide or death from any cause. Kaplan-Meier methods will used.
Time Frame: From date of study entry until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 58 months.
Population: All participants who started therapy
Measure: Count of Participants; unit: Participants
Arm/Group | KRdD Followed by Auto-HCT | KRdD Only
Number analyzed (Participants) | 123 | 0
Participants | 90 |

8. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from date of study enrollment until death from any cause.
Time Frame: as for outcome 7
Population: All participants who started therapy
Measure: Count of Participants; unit: Participants
Arm/Group | KRdD Followed by Auto-HCT | KRdD Only
Number analyzed (Participants) | 123 | 0
Participants | 108 |

ADVERSE EVENTS:
Time Frame: 5 years
Description: Risk of zero relates to arm that did not have enrollment since all participants were transplant eligible
Arm/Group | KRdD Followed by Auto-HCT | KRdD Only
All-Cause Mortality (participants affected / at risk) | 15/123 | 0/0
Serious Adverse Events (participants affected / at risk) | 14/123 | 0/0
Other Adverse Events (participants affected / at risk) | 123/123 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KRdD Followed by Auto-HCT (N=123) | KRdD Only (N=0)
Lung Infection (Infections and infestations) | 8 (8) | 0 (0)
Thomboembolism (Vascular disorders) | 3 (3) | 0 (0)
sudden death (Cardiac disorders) | 2 (2) | 0 (0)
Viral pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KRdD Followed by Auto-HCT (N=123) | KRdD Only (N=0)
Neutropenia (Blood and lymphatic system disorders) | 51 (51) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 34 (34) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 23 (23) | 0 (0)
fatigue (General disorders) | 69 (69) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 68 (68) | 0 (0)
maculopapular rash (Skin and subcutaneous tissue disorders) | 50 (50) | 0 (0)
Nausea (Gastrointestinal disorders) | 49 (49) | 0 (0)
constipation (Gastrointestinal disorders) | 48 (48) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 45 (45) | 0 (0)
diarrhea (Gastrointestinal disorders) | 43 (43) | 0 (0)
insomnia (General disorders) | 35 (35) | 0 (0)
infusion-related reaction (General disorders) | 34 (34) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 34 (34) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 33 (33) | 0 (0)
hypertension (Vascular disorders) | 32 (32) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT03224507/Prot_SAP_001.pdf